CLINICAL TRIAL: NCT06434168
Title: A Pilot and Feasibility Study of a Yoga Intervention in Heart Failure Patients With Mild Cognitive Impairment
Brief Title: Impact of Yoga on Cognitive Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: VCOM, Auburn campus (Unknown)
Responsible Party: Principal Investigator, Chin-Yen Lin, Assistant Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AU-24-001
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Mild Cognitive Impairment
Keywords: Yoga intervention; cognitive function
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga intervention (Experimental)
  Interventions: Behavioral: Yoga intervention
- Control condition (Placebo Comparator)
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: Yoga intervention — Patients in the yoga group will receive a 60-minute session, twice per week over 12 weeks for a total of 24 sessions. Each yoga session consists of a warm-up, yoga postures standing or seated depending on the capability of the patient, and relaxation.
  Arms: Yoga intervention
Behavioral: Control condition — Patients in the control group will receive care-as-usual from their healthcare providers and will be asked to avoid engaging in yoga during their 3 months in the study.
  Arms: Control condition

SUMMARY:
Mild cognitive impairment is highly prevalent in patients with heart failure and results in poor well-being and quality of life. While yoga has proven effective in promoting cognitive health in older adults through its gentle movements, controlled breathing, and meditation, its effects on patients with heart failure remain unknown. Therefore, this feasibility and pilot study plans to deliver a 12-week yoga intervention and test its effects on cognitive function in patients with heart failure and mild cognitive impairment.

DETAILED DESCRIPTION:
A prospective, 2-arm comparative feasibility design will be used. The investigators will enroll 24 patients with a confirmed heart failure diagnosis with mild cognitive impairment. Patients will be randomized equally into yoga intervention or control group. Patients in the yoga intervention group will receive a 60-minute yoga session twice per week for 12-week. Survey, cognitive function data, MRI scans, and blood samples will be collected at baseline and at 3 months (after completion of yoga intervention).

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 years and older
* Confirmed heart failure diagnosis with mild cognitive impairment
* New York Heart Association functional class II-IV

Exclusion Criteria:

* Co-existing neurological disorders, traumatic brain injury, psychiatric disorders, or terminal illnesses
* Have implanted defibrillator, left ventricular assist device placement or cardiac transplant
* Have any other implanted metals that interfere with the MRI magnetic field for patient safety
* Substance abuse
* Pregnant
* Unable to perform yoga due to physical limitations or severity of illness

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain structure | Change from 0-12 weeks, from baseline pre-intervention to 12 weeks post-intervention
  Using structural magnetic resonance imaging to examine brain structure between intervention and control groups. Less brain alteration is optimal.
Brain functional connectivity | Change from 0-12 weeks, from baseline pre-intervention to 12 weeks post-intervention
  Functional magnetic resonance imaging is used to examine functional connectivity between intervention and control groups. A balance of activity across different brain regions is optimal.
Cognitive function | Change from 0-12 weeks, from baseline pre-intervention to 12 weeks post-intervention
  Using cognitive tests to examine cognitive function and performance between intervention and control groups. A higher score on cognitive tests indicates better cognitive function.
Serum brain-derived neurotrophic factor | Change from 0-12 weeks, from baseline pre-intervention to 12 weeks post-intervention
  A blood sample will be obtained using phlebotomy to measure the levels of serum brain-derived neurotrophic factor and reported in pg/mL. Higher concentrations are optimal.

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No